CLINICAL TRIAL: NCT06833034
Title: To Compare the Effectiveness of a Novel Closed Exposure Technique With Removal of Bone Tissue and a Conventional Technique During Treatment of Palatally Impacted Maxillary Canines by Closed Surgical Exposure and Fixed Orthodontic Appliance
Brief Title: Comparing a Novel Closed Exposure Technique to a Conventional Method for Palatally Impacted Maxillary Canines
Acronym: PDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Ortodontilund AB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dnr 2023-02596-02
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Impacted Canines
Keywords: impacted maxillary canines

STUDY DESIGN:
Intervention Model Description: Surgical technique After anesthesia and rising of the mucoperiosteal flap the patients are randomized, by a staff member not involved in the study, for further treatment into one of two groups: A) The conventional surgical procedure without additional bone removal and B) the novel surgical procedure with additional bone removal.
  In the end of the surgical session, the auxiliary attachment is placed on the crown of the canine and the incision is made on the palatal flap letting the chain protrude exactly where the canine is placed.
  The flap is then sutured with conventional sutures and the patients are instructed to rinse with Chlorhexidine until the sutures are removed after 10 days at the orthodontic clinic and the chain is activated and followed as normal procedure in the orthodontic treatment.
  The surgery will be performed by one surgeon. The orthodontic treatment will be performed by four orthodontists at the three orthodontic clinics.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional surgical method (Active Comparator): The conventional surgical method usually used in the clinic
  Interventions: Procedure: The novel surgical method
- The novel surgical method (Experimental): Additional bone removal in intendet direction of tooth movement
  Interventions: Procedure: The conventional surgical method

INTERVENTIONS:
Procedure: The novel surgical method — Additional bone removal in intended direction for tooth movement
  Arms: The conventional surgical method
Procedure: The conventional surgical method — The conventional method to use surgery
  Arms: The novel surgical method

SUMMARY:
A multi-center Randomized Clinical Trial, (RCT) on treatment effectiveness of two different closed surgical exposure techniques, one including additional bone removal and a second conventional without removal of additional bone, during treatment of palatally impacted maxillary canines.

A comparison between the two methods regarding the anchorage situation for the incisors will be performed as well.

Introduction Surgical exposure of impacted maxillary canines together with orthodontic treatment has long been advocated. Closed exposure with placement of an auxiliary attachment with a chain, followed by traction of the canine with orthodontic forces is commonly clinical used to avoid complications with the open procedure (Kokich 2004). Both open and closed methods and orthodontic treatment are one of the most time-consuming orthodontic treatments. Therefore, it is valuable to try to find methods which can reduce the total treatment time and make the treatments as comfortable as possible for the patient.

To reduce the treatment time, study I investigates a novel strategy for traction of the canine. Another strategy to reduce the treatment time might be to facilitate the movement of the canine by additional bone removal in the eruption direction out to the alveolar crest. This has been used of a few orthodontists in one clinic for some years. No negative side-effects have been seen. There are, however, no studies for comparison of the two techniques.

Aim The primary aims of this Randomized Clinical Trial (RCT) is to evaluate the treatment effectiveness of two different surgical closed exposure techniques of palatally impacted canines before the orthodontic treatment; a) with removal of bone in traction direction and b) without removal of bone in traction direction and to evaluate the anchorage situations.

Outcome variables The outcome variables will be: 1) Treatment time for the canine to be exposed in the oral cavity; 2) Treatment time for the canine to be in the dental arch and 3) Treatment time for the canine to have reached the right position in the dental arch.

Subjects Sixty-six patients between 10-18- years, will be recruited to the study. Patients with palatally impacted maxillary canines are consecutively recruited at three orthodontic clinics in Lund, Karlshamn and Ängelholm.

DETAILED DESCRIPTION:
Study Title: Comparing Novel and Conventional Techniques for Treating Palatally Impacted Maxillary Canines

Study Overview: This clinical study aims to compare the effectiveness and patient experiences of two different techniques used to treat palatally impacted maxillary canines. These are teeth that have not properly emerged into the mouth and are instead located in the palate. The study will focus on two specific techniques: a novel closed exposure technique that involves the removal of bone tissue, and a conventional traction technique.

Study Objectives:

Effectiveness and Patient Experience: The primary goal is to evaluate and compare the effectiveness of the novel and conventional techniques in treating palatally impacted maxillary canines. Additionally, the study will assess patient experiences, particularly focusing on pain and discomfort during the treatment process.

Anchorage Situation: The study will also compare the anchorage situation for the incisors (front teeth) when using the novel closed exposure technique versus the conventional technique.

Study Methods: Participants in the study will undergo treatment for their palatally impacted maxillary canines using either the novel closed exposure technique or the conventional traction technique. Both techniques involve closed surgical exposure and the use of fixed orthodontic appliances. Detailed descriptions of both techniques will be provided to ensure a clear understanding of the procedures.

Expected Outcomes: The study aims to determine which technique is more effective in treating palatally impacted maxillary canines and to understand the patient experiences associated with each technique. By comparing the two methods, the study hopes to provide valuable insights into the best practices for treating this dental condition.

Significance: Palatally impacted maxillary canines can cause significant dental issues if not properly treated. This study will contribute to the field of orthodontics by providing evidence-based recommendations for the most effective and comfortable treatment methods. The findings will help dental professionals make informed decisions and improve patient care.

ELIGIBILITY:
Inclusion Criteria:

• Patients with palatally impacted maxillary canine on one side, in sector 2-4 and with angle <45º are included.

Exclusion Criteria:

* Patients with clefts or syndromes
* Patients with earlier orthodontic treatment
* Patients with canines with angle >45º (fig.1)
* Patients with canines with impacted canines in sectors 1 or 2

Ages: 10 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Treatment time for the canine to be exposed in the oral cavity | 24 months
  The primary outcome measure for this study is the treatment time required for the palatally impacted maxillary canine to be exposed in the oral cavity. This will be measured in months from the start of the treatment until the canine is visible.

SECONDARY OUTCOMES:
Treatment time for the canine to align and reach its final position | 24 months
  Secondary outcome measures include the treatment time for the canine to align within the dental arch and the time to reach its final position within the dental arch. This will be measured in months from the start of the treatment.

OTHER OUTCOMES:
Patient-reported pain and discomfort | 24 months
  Patient-reported outcomes such as pain and discomfort during the treatment process will also be assessed using standardized questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sonesson, Docent, Study Director — Malmö University
Locations (2):
- Sweden (2):
  - Borgska villans specialisttandvård, Lund, Skåne County
  - Malmö universitet, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No